CLINICAL TRIAL: NCT02115048
Title: A Randomized Open-label Phase II Study of Letrozole Plus Afatinib Versus Letrozole Alone in First-line Treatment of Advanced ER+, HER2- Postmenopausal Breast Cancer With Low ER Expression
Brief Title: Clinical Study for the Treatment of Breast Cancer: the Patient Will Receive Afatinib Plus Letrozole or Letrozole Alone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was completed as per amended protocol. Protocol was amended to close enrollment earlier than initially planned (study continued as per plan).
Sponsor: Translational Research in Oncology (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIO 020
Record Dates: First submitted 2014-04-09; First posted 2014-04-15 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Continuous regimen of oral Letrozole 2.5 mg daily
  Interventions: Drug: Letrozole
- Arm B (Experimental): Continuous regimen of oral Letrozole 2.5 mg daily plus oral Afatinib 30 mg daily
  Interventions: Drug: Letrozole; Drug: Afatinib

INTERVENTIONS:
Drug: Letrozole
Drug: Afatinib
  Arms: Arm B

SUMMARY:
The purpose of the study is to compare the efficacy of treatment with afatinib plus letrozole to treatment with letrozole alone in women diagnosed with a specific type of breast cancer.

DETAILED DESCRIPTION:
This is an open-label, multicenter, international, randomized, Phase II clinical trial that will assess the efficacy and safety of letrozole in combination with afatinib(oral epidermal growth factor receptor (EGFR ) inhibitor) versus letrozole monotherapy for the first-line treatment of postmenopausal women with ER+, Human Epidermal Growth Factor Receptor 2 (HER2) negative advanced breast cancer with low ER expression.

In order to assess the level of estrogen receptor (ER) expression we will use a semi-quantitative scoring system (McClelland, 1990) defined as :

H-score = (% of cells stained at intensity category 1x1) + (% of cells stained at intensity category 2x2) + (% of cells stained at intensity category 3x3).

This formula results in an H-score in the range of 0-300 where 300 equals 100% of tumor cells stained strongly (i.e., 3+). Low ER expression will be defined as tumor sample with H-score below 160 (Finn, 2009).

All subjects who consented for the study must submit a tumor sample to the designated central laboratory for central confirmation of ER / Progesterone receptor (PR) and HER2 statuses and determination of the H-score. This will be assessed prior to randomization.

Subjects with HER2 negative, ER+ advanced breast cancer with low ER expression defined as H-score between 1 and 159 will enter screening phase and perform the required screening assessments.

Eligible subjects will be randomly assigned in a 1:1 ratio and stratified according to sites of disease (bone only disease vs. other) and prior administration of hormonal therapy in neo/adjuvant setting (Yes vs. No) to either:

Arm A : Continuous regimen of oral letrozole 2.5 mg until progression of disease or any other study treatment discontinuation criteria.

or Arm B : Continuous regimen of oral letrozole 2.5 mg daily plus oral afatinib 30 mg daily until progression of disease or any other study treatment discontinuation criteria.

IN ADDITION the following applies whichever comes first:

* If the patients treated with the combination of afatinib and letrozole (arm B) discontinue the trial treatment (whatever the reason) before 30 November 2018, the patients from the other arm (arm A, letrozole alone) still on treatment will also be discontinued from the trial at the same time. They may continue receiving letrozole using commercial drug as standard of care according to their treating physician discretion.
* If the patients treated with afatinib and letrozole (arm B) have not discontinued the trial treatment by 30 November 2018, all patients currently on treatment in the trial (including the ones only treated by letrozole alone (arm A)) will be discontinued from the trial at that time. They may continue receiving their treatment if in alignment with their treating physician judgment as follows:
* Patients in arm A: may continue receiving letrozole using commercial drug as standard of care according to their treating physician discretion.
* Patients in arm B: may continue receiving afatinib in the context of alternative drug supply outside the clinical trial as appropriate according to local legislation. Additionally, they may continue receiving letrozole using commercial drug as standard of care according to their treating physician discretion.

Once the patient is discontinued from trial treatment and has undergone the End of Treatment Visit, she will be permanently discontinued from the trial and treated as per local clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Postmenopausal females, 18 years of age or older.
* Histologically or cytologically proven diagnosis of adenocarcinoma of the breast with evidence of locally recurrent disease not amenable to resection or radiation therapy with curative intent, or metastatic disease.
* HER2 negative breast cancer. Central testing (required for all subjects) must demonstrate that the tumor is HER2 negative by FISH or Immunohistochemistry (IHC).
* ER positive breast cancer. Central testing (required for all subjects) must demonstrate that the tumor is ER+ with low expression (H-score [1-159]).
* Paraffin-embedded tumor block(s) or 15 to 20 unstained slides available for centralized assessment of ER, PR, and HER2.
* Measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 or bone-only non measurable disease.
* Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1.
* Adequate hematological, hepatic and renal functions.
* Baseline left ventricular ejection fraction (LVEF) 50%.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease.
* Prior treatment with any type of systemic therapy for advanced disease.
* Prior treatment with letrozole in (neo)adjuvant setting with disease-free interval ≤ 12 months from completion of treatment until randomization.
* Prior treatment with any anti HER-family targeted therapy in (neo)adjuvant setting.
* Any concurrent or previous malignancy within 5 years prior to randomization, except for adequately and radically treated basal or squamous skin cancer, or carcinoma in situ of the cervix, or other non-invasive/in-situ neoplasm.
* Non-measurable disease according to RECIST 1.1, with the exception of bone-only non-measurable disease.
* Known pre-existing interstitial lung disease.
* Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom.
* History or presence of clinically relevant cardiovascular abnormalities as per investigator assessment.
* Any other concomitant serious illness or organ system dysfunction as per investigator assessment
* Any contraindication to oral agents.
* Active hepatitis B infection, active hepatitis C infection or known HIV carrier.
* Known or suspected active drug or alcohol abuse.
* Known hypersensitivity to afatinib or letrozole or the excipients of any of the trial drugs.
* Concomitant treatment with strong inhibitor of P-gp.
* Any ongoing acute clinically significant toxic effect of prior anticancer therapy or any persisting complication of prior surgery.
* Subjects with known history of keratitis, ulcerative keratitis or severe dry eye.
* Participation in the active phase of other clinical trials of investigational agents in which last study treatment was administered within 2 weeks prior to randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-07; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finn, MD, Study Chair — University of California, Los Angeles
Locations (26):
- United States (9):
  - St. Jude Heritage Healthcare, Fullerton, California
  - University of California Los Angeles Hematology Oncology, Los Angeles, California
  - West Valley Hematology Oncology Medical Group, Northridge, California
  - DBA Torrance Memorial Physician Network/Cancer Care Associates, Redondo Beach, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Orlando Health, Inc., Orlando, Florida
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hope Women's Cancer Centers, Asheville, North Carolina
- Bosnia and Herzegovina (3):
  - University Hospital Clinical Center Banja Luka, Oncology Clinic, Banja Luka
  - Clinical Center of University in Sarajevo, Clinic for Oncology, Sarajevo
  - University Clinical Center Tuzla Clinic for Oncology, Hematology and Radiotherapy, Tuzla
- Romania (6):
  - Filantropia Clinical Hospital, Bucharest
  - County Emergency Clinical Hospital Cluj-Napoca Oncology Department, Cluj-Napoca
  - SC Medisprof SRL, Cluj-Napoca
  - County Hospital Ploiesti, Ploieşti
  - County Emergency Hospital "Sf Ioan cel Nou", Suceava
  - Oncomed SRL Timisoara, Timișoara
- Spain (8):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de Especialidades de Jerez de La Frontera, Jerez de la Frontera
  - Hospital Clínico Universitario Virgen de La Arrixaca, Murcia
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitari de Sant Joan de Reus, Reus
  - Hospital Universitario Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For all patients consented on the trial, a tumor sample was sent to the central lab for testing of ER/PR and HER2 and determination of the H-score. This was assessed prior to randomization. Patients with HER2 negative, ER+ advanced breast cancer with low ER expression defined as H-score between 1 and 159 entered screening phase.
Groups:
- Arm A: Letrozole 2.5 mg
- Arm B: Letrozole 2.5 mg + Afatinib 30 mg
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 23 | 21
Completed (Trial terminated early and only 44 patients enrolled, preventing appropriate statistical calculation) | 23 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 44 patients were enrolled in the trial; 23 in Arm A and 21 in Arm B. All patients started and completed treatment at the time of reporting.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 9 | 11 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Romania | 3 | 5 | 8
  United States | 9 | 6 | 15
  Bosnia and Herzegovina | 4 | 3 | 7
  Spain | 7 | 7 | 14
Menopausal Status [Count of Participants; unit: Participants]
  Pre-Menopausal | 0 | 0 | 0
  Post-Menopausal | 23 | 21 | 44
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG Scale of Performance Status is a measurement used to describe a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.).
  Patients with ECOG 0 are in better general condition than patients with ECOG 1:
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    0 | 12 | 14 | 26
    1 | 11 | 7 | 18
Weight (kg) [Mean (Standard Deviation); unit: kg] — Weight measured in kg.
  kg | 77.39 (16.25) | 69.59 (11.14) | 73.67 (14.44)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the time from randomization until date of progression (assessed by Response Evaluation Criteria in Solid Tumors - RECIST) or death due to any cause, whichever occurs first. For evaluation of PFS, the randomization date for each patient was the "start date". If the status at the last assessment date was "Non-complete response/ Non-progressive disease" or "Complete response", then the patient was considered "censored". If the status at the last assessment for any tumor was "Progressive disease", then the patient was considered as having an event.
  Progressive disease is defined using RECIST v1 .1 as a ≥ 20% increase in the sum of the longest diameter of target lesions compared with the smallest-sum longest diameter recorded or the appearance of one or more target or non-target new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Tumor assessments were every 12 weeks up to 9 months (average) for subjects in Arm A or up to 14 months (average) for subjects in Arm B.
Population: The timeframe specifies when tumor assessments were performed. Enrollment was closed prematurely due to low recruitment (only 44 participants enrolled) compared to what was initially planned (150 participants), therefore no statistical evaluations were completed (including PFS).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 18
Participants
  Failed (Progressed or Died) | 4 | 2
  Censored | 14 | 16

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time from randomization until death to any cause.
  For subjects in which treatment is discontinued for reasons different than Progression Disease: after treatment and up to documentation of disease progression: Overall Survival is assessed every 12 weeks
Time Frame: Under treatment: every 4 wks up to 9 months (average) for subject in the Arm A or up to 14 months (average) for subjects in Arm B. After documentation of disease progression up to the end of the study: every 6 months up to 42 months
Population: The timeframe specifies when tumor assessments were performed. Enrollment was closed prematurely due to low recruitment (only 44 participants enrolled) compared to what was initially planned (150 participants), therefore no statistical evaluations were completed (including OS).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 18
Participants
  Died | 2 | 0
  Censored | 16 | 18

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the proportion of randomized subjects achieving a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST). As per RECIST (version 1.1):
  CR is defined as disappearance of all target and non target lesions - lymph node (LN) <10mm.
  PR is defined as at least a 30% decrease in the Sum of Diameters, taking as reference the Baseline Sum of Diameters
Time Frame: Tumor assessment: every 12 weeks up to 9 months (average) for subjects in Arm A or up to 14 months (average) for subjects in Arm B.
Population: The timeframe specifies when tumor assessments were performed. Enrollment was closed prematurely due to low recruitment (only 44 participants enrolled) compared to what was initially planned (150 participants), therefore no statistical evaluations were completed (including ORR).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 18
Participants
  Complete Response (CR) | 2 | 1
  Death | 2 | 0
  Progessive Disease (PD) | 2 | 2
  Non-CR / Non-PD | 12 | 15

4. Secondary Outcome: Time to Tumor Progression (TTP)
Description: As per Response Evaluation Criteria In Solid Tumors (RECIST). Time to progression (TTP) is defined as the time interval from date of randomization to date of the first documented objective tumor progression.
Time Frame: Tumor assessments: every 12 weeks up to 9 months (average) for subjects in Arm A or up to 14 months (average) for subjects in Arm B.
Population: The timeframe specifies when tumor assessments were performed. Enrollment was closed prematurely due to low recruitment (only 44 participants enrolled) compared to what was initially planned (150 participants), therefore data for TTP was not produced due to the small number of patients (evaluation would not produce meaningful data).
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Participants who experienced at least one Treatment Emergent Adverse Event (TEAE) are presented. Participants with at least one serious TEAE, those who had at least one TEAE related to letrozole or afatinib (serious/non-serious), including participants who experienced a grade 3/4 TEAE, or who discontinued/died as a result of their TEAE are listed by treatment arm. Adverse events were tabulated by system organ class, preferred term and toxicity grade by treatment arm. For subjects in which treatment was discontinued for reasons different than progression of disease, the assessment was conducted every 12 weeks following treatment, and up to documentation of disease progression.
  ** Enrollment was closed prematurely due to low recruitment (only 44 participants enrolled) compared to what was initially planned (150 participants), therefore no statistical evaluations were completed. Adverse event data collected are described per arm but no statistical comparison was made.
Time Frame: Under treatment: every 4 wks up to 9 months (average) for subjects in Arm A or up to 14 months (average) for subjects in Arm B. After documentation of disease progression up to the end of the study: every 6 months up to 42 months
Population: Participants who experienced at least one Treatment Emergent Adverse Event (TEAE) are listed. Participants with at least one serious TEAE, those who had at least one TEAE related to letrozole or afatinib (serious/non-serious), including participants who experienced a grade 3/4 TEAE, or who discontinued/died as a result of their TEAE are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 23 | 21
Participants
  Patient having at least one TEAE | 16 | 20
  Patient having at least one serious TEAE | 5 | 2
  At least one TEAE related to letrozole | 6 | 11
  At least one TEAE related to afatinib | 0 | 18
  At least one serious TEAE related to letrozole | 0 | 0
  At least one serious TEAE related to afatinib | 0 | 1
  Patient having at least one grade 3/4 TEAE | 7 | 3
  TEAE leading to discontinuation - letrozole | 1 | 1
  TEAE leading to discontinuation - afatinib | 0 | 1
  Fatal TEAE | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years, 3 months (28 August 2014 to 30 November 2018). 28 August 2004 corresponds to the first enrolment in the trial, and 30 November 2018 corresponds to the 'end of data' collection period. All participants were assessed for adverse events (AEs) from their date of enrolment to the end of the observation period, which as per protocol is defined as 30 days following their last treatment intake - during this time serious AEs also had to be reported.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 2/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 5/23 | 2/21
Other Adverse Events (participants affected / at risk) | 16/23 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=23) | Arm B (N=21)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=23) | Arm B (N=21)
Diarrhoea (Gastrointestinal disorders) | 2 | 15
Nausea (Gastrointestinal disorders) | 3 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 6
Abdominal Distension (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 1 | 6
Paronychia (Infections and infestations) | 0 | 6
Urinary Tract Infection (Infections and infestations) | 0 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 1
Weight Increased (Investigations) | 2 | 4
Weight Decreased (Investigations) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 6
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 5
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
Enrolment was closed prematurely with only 44 participants enrolled compared to what was initially planned (150 participants). Thus, preventing appropriate statistical evaluation (primary/secondary objectives no longer applicable as per protocol).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication, abstract or presentation of the Study will be made without the approval of the Study Steering Committee (SCC). The SSC will be solely responsible for the analysis, interpretation and public disclosure of the results of the trial in accordance with the statistical plan.

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT02115048/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT02115048/SAP_001.pdf